CLINICAL TRIAL: NCT05172180
Title: Correction of Metabolic Disorders and Its Effect on Respiratory Function of Lungs in Patients With Severe COVID-19
Acronym: CARECOVID
Status: Completed | Type: Observational
Sponsor: POLYSAN Scientific & Technological Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Other Study IDs: CARECOVID
Record Dates: First submitted 2021-12-20; First posted 2021-12-29 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2023-12

CONDITIONS: COVID-19
Keywords: COVID-19; METABOLIC DISORDERS; Respiratory function of the lungs
MeSH Terms: conditions — COVID-19; Metabolic Diseases | interventions — Reamberin; Ringer's Solution

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The control group: The control group consisted of 54 patients who received Ringer's solution at an average daily dose of 8.1 ml/kg/day as the main infusion solution from the time of transfer to the intensive care unit
  Interventions: Drug: Ringer's solution
- The test group: Fifty one patients in the test group received the balanced succinate-containing crystalloid solution Reamberin (meglumine sodium succinate) at an average daily dose of 8.3 ml/kg/day for the same purpose
  Interventions: Drug: Reamberin

INTERVENTIONS:
Drug: Reamberin — the balanced succinate-containing crystalloid solution Reamberin (meglumine sodium succinate)
  Groups: The test group
Drug: Ringer's solution — Ringer's solution at an average daily dose of 8.1 ml/kg/day
  Groups: The control group

SUMMARY:
Objective of the study: to investigate the effect of meglumine succinate solution on the dynamics of metabolic blood parameters and respiratory function of the lungs in intensive care patients with new coronavirus infection. An observational prospective study included 105 patients with a severe course of novel coronavirus infection

ELIGIBILITY:
Inclusion Criteria:

1. age 18-70 years;
2. diagnosis of SARS-COV-2 NCI confirmed by laboratory tests;
3. the lung lesion volume on CT scan is significant or subtotal - CT 3-4;
4. initiation of infusion therapy on the 1st day after patient admission to ICU

Exclusion Criteria:

* 1) presence of initial indications for transfer to invasive ALV at the time of screening; 2) history of Reamberin intolerance; 3) administration of other polyelectrolyte solutions with reserve alkalinity carriers; 4) pregnancy and postpartum; 5) severe renal failure requiring renal replacement therapy; 6) severe hepatic failure (Child-Pugh class C or higher); 7) diabetes mellitus; 8) terminal stage of other chronic incurable diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe novel coronavirus infection COVID-19 (NCI) who were treated at the intensive care unit (ICU)
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Mortality, % | from date of treatment start until the date of death or the date of discharge from hospital
  Proportion of patients died during the period of hospital stay
Duration of treatment at ICU, days | from date of treatment start until the date of death or the date of discharge from hospital
  Duration of treatment at ICU
Duration of treatment after ICU, days | from date of treatment start until the date of death or the date of discharge from hospital
  Duration of treatment after ICU

SECONDARY OUTCOMES:
Glucose | baseline, day 2, day 3, day 5, day 11
  Venous blood Glucose
Lactate | baseline, day 2, day 3, day 5, day 11
  Venous blood Lactate
pH | baseline, day 2, day 3, day 5, day 11
  Blood gases
BE | baseline, day 2, day 3, day 5, day 11
  Blood gases
Dynamics of right diaphragm excursion, cm | baseline, day 2, day 3, day 5, day 11
  Diaphragm mobility
Total duration of inpatient treatment, days | from date of treatment start until the date of death or the date of discharge from hospital
  Total duration of inpatient treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Nizhegorodskaya Regional Clinical Hospital named after N.A. Semashko, Nizhny Novgorod, Russia

REFERENCES:
- See also: Metabolic therapy and its impact on lung respiratory function in patients with severe COVID-19 A.Yu. Yakovlev, A.A. Pevnev, M.V. Dudorova, Yu.V. Ilyin, M.S. Belous https://doi.org/10.17816/KMJ2022-364 — https://kazanmedjournal.ru/kazanmedj/article/view/100007